CLINICAL TRIAL: NCT01605708
Title: Randomized, Double-Blind, Placebo-Controlled, Sequential Ascending Dose Study of the Clinical Activity, Safety, Tolerability and Pharmacokinetics of a Single IV Dose of REGN846 in Refractory Moderate-to-Severe Pruritus in Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study to Assess the Clinical Activity of a Sequential Dose of REGN846 on Refractory Pruritus in Patients With Atopic Dermatitis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R846-AD-1105
Record Dates: First submitted 2011-10-12; First posted 2012-05-25 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-05

CONDITIONS: Pruritus; Atopic Dermatitis
Keywords: Itching
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 1 (Experimental)
  Interventions: Drug: REGN846

INTERVENTIONS:
Drug: REGN846 — Dose 1

SUMMARY:
The purpose of this study is to assess the clinical activity on refractory moderate-to-severe pruritus of a single intravenous (IV) dose of REGN846 in adult patients with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria include, but are not limited to the following:

1. Men and women between the ages of 18 and 65; women must be postmenopausal or surgically sterile
2. Patients must have applied a stable dose of an additive-free, basic, bland emollient twice daily for at least 7 days before the baseline visit
3. Chronic Atopic Dermatitis (AD)
4. Body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive.
5. Refractory pruritus for ≥ 6 weeks before screening. Pruritus should be associated only with AD and not with any other condition(s).
6. Itching associated with AD

Exclusion Criteria:

Exclusion criteria include, but are not limited to the following:

1. A history of listeriosis.
2. Presence of any 1 of the following tuberculosis (TB) criteria:

   1. A history of active TB
   2. A positive QuantiFERON TB test at the screening visit
   3. Chest radiograph (posterior-anterior and lateral views) at screening or within 3 months before the screening visit (radiology report must be available) with results consistent with prior TB infection (including but not limited to apical scarring, apical fibrosis, or multiple calcified granuloma). This does not include non-caseating granulomata.
3. Persistent chronic or active recurring infection requiring treatment with antibiotics, antivirals, or antifungals within 4 weeks prior to the screening visit.
4. Any clinically significant physical abnormalities observed during the screening visit.
5. Diabetic, hypertensive, or any known atherosclerotic vascular disease.
6. Hospitalization for any reason within 60 days of the screening visit.
7. History of or positive human immunodeficiency virus (HIV) screen result at the screening visit.
8. History of positive blood test for hepatitis B/hepatitis C or positive hepatitis screen result at the screening visit.
9. Known sensitivity to doxycycline or tetracycline.
10. Known sensitivity to any of the components or excipients of the investigational product formulation or history of hypersensitivity to any biologic agent.
11. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer), of the investigational drug prior to the screening visit.
12. Any medical or psychiatric condition that in the opinion of the investigator or Regeneron, would place the patient at risk, interfere with participation in the study or interfere with the interpretation of study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Clinical Activity | Week 2
  To assess the clinical activity on refractory moderate-to-severe pruritus of a single intravenous (IV) dose of REGN846 in adult patients with moderate-to-severe AD.
Clinical Activity | Week 4
  To assess the clinical activity on refractory moderate-to-severe pruritus of a single intravenous (IV) dose of REGN846 in adult patients with moderate-to-severe AD.
Clinical Activity | Week 6
  To assess the clinical activity on refractory moderate-to-severe pruritus of a single intravenous (IV) dose of REGN846 in adult patients with moderate-to-severe AD.

SECONDARY OUTCOMES:
Safety and tolerability a single IV dose of REGN846 | Week 1 - Week 6
  To assess the safety and tolerability of REGN846 in adult patients who have moderate-to-severe AD with refractory moderate-to-severe pruritus.
Pharmacokinetic (PK) profile of a single IV dose of REGN846 | Week 1 - Week 6
  To assess the PK profile of REGN846 in adult patients who have moderate-to-severe AD with refractory moderate-to-severe pruritus.
Immunogenicity of a single IV dose of REGN846 | Week 1 - Week 6
  To assess the immunogenicity of REGN846 in adult patients who have moderate-to-severe AD with refractory moderate-to-severe pruritus.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (14):
- Finland (2):
  - Helsinki
  - Tampere
- Germany (8):
  - Berlin
  - Dresden
  - Erfurt
  - Frankfurt
  - Mahlow
  - Mainz
  - Osnabrück
  - Tübingen
- Poland (4):
  - Bydgoszcz
  - Poznan
  - Warsaw
  - Wroclaw